CLINICAL TRIAL: NCT04275505
Title: Efficacy of Shortwave Diathermy in Ulnar Nerve Entrapment on the Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: naciyebilginbadur
Record Dates: First submitted 2020-02-13; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Ulnar Nerve Entrapment at Elbow
Keywords: shortwave diathermy, ulnar nerve entrapment at elbow
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: this study has 2 groups of participants. treatment group and control group. It is designed as randomized controlled double blind clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the participants did not know if they were in tratment group or control group. both of the group participants were asked to put their elbow into the shortwave diathermy device and they did not know if the device was turned on or off.
  the investigator (Naciye Bilgin Badur) did not know the participants group while performing physical examination before and after intervention in control visits.
  investigator and outcome assessor are the same person who is Naciye Blgin Badur

ARMS (2):
- treatment group (Active Comparator): the participants were given 10 sessions of shortwave diathermy treatment and elbow splint and told to avoid symptom provoking activities
  Interventions: Other: shortwave diathermy treatment
- control group (Placebo Comparator): the participants were given 10 sessions of placebo shortwave diathermy treatment (the device was not turned on), elbow splint and told to avoid symtpom provoking activities
  Interventions: Other: placebo shortwave diathermy treatment

INTERVENTIONS:
Other: shortwave diathermy treatment — shortwave diathermy is a deep heating physical therapy agent. It was found efficiaous in carpal tunnel syndrome which is an entrapment neuropathy like ulnar nerve entrapment so it was hypothesised that shortwave diathermy could be an effective treatment method in ulnar nerve entrapment.
  Arms: treatment group
Other: placebo shortwave diathermy treatment — shortwave device was not turned on while participants were asked to put their elbow into the device
  Arms: control group

SUMMARY:
It was aimed to see if there is any efficacy of short wave diathermy (SWD) in the treatment of ulnar nerve entrapment at the elbow (UNE). Ulnar nerve entrapment, following carpal tunnel syndrome (CTS), is the second most common upper extremity entrapment neuropathy. Ulnar nerve is compressed mostly in elbow region because of its anatomy. Conservative treatment choices are limited in ulnar nerve entrapment neuropathy and very few studies about UNE, are available in literature.

The aim of this study was researching the efficacy of SWD which is a deep heating modality in treatment of UNE. SWD is used either continuous or pulsed mode. Continuous SWD is used for the purpose of heating.

MATERIALS AND METHODS: 61 adult patients, who had been diagnosed with UNE clinically and electrophysiologically, were randomly assigned into two groups. Ten sessions of SWD was applied to the patients in the treatment group as 5 sessions per week for 2 weeks. Ten sessions of placebo SWD was applied to the patients in the control group as 5 times a week, for 2 weeks. All patients in both groups were given elbow splints and were informed to avoid symptom provocating activities. Patients were evaluated at baseline, at the end of the treatment and,1 and 3 months after the treatment. Besides physical examination, quick-DASH (disabilities of arm, shoulder, hand) and SF-36 were used to evaluate activities of daily life, dynamometer was used to evaluate grip force and VAS was used to evaluate pain severity.

DETAILED DESCRIPTION:
efficacy of short wave diathermy in ulnar nerve entrapment on the elbow

ABSTRACT

OBJECTIVE: Efficacy of short wave diathermy (SWD) in the treatment of ulnar nerve entrapment at the elbow (UNE).

MATERIALS AND METHODS: 61 adult patients, who had been diagnosed with UNE clinically and electrophysiologically, were randomly assigned into two groups. Ten sessions of SWD was applied to the patients in the treatment group as 5 sessions per week for 2 weeks. Ten sessions of placebo SWD was applied to the patients in the control group as 5 times a week, for 2 weeks. All patients in both groups were given elbow splints and were informed to avoid symptom provocating activities. Patients were evaluated at baseline, at the end of the treatment and,1 and 3 months after the treatment. Besides physical examination, quick-DASH (disabilities of arm, shoulder, hand) and SF-36 were used to evaluate activities of daily life, dynamometer was used to evaluate grip force and VAS was used to evaluate pain severity.

INTRODUCTION

Ulnar nerve entrapment, following carpal tunnel syndrome (CTS), is the second most common upper extremity entrapment neuropathy. Ulnar nerve is compressed mostly in elbow region because of its anatomy. Ulnar nerve entrapment neuropathy diagnosis depends on symptoms, physical examination and electrodiagnostical tests (1). The incidence of ulnar nerve entrapment in elbow (UNE) was found as 25.2/100000 in Siena, a district of Italy (2). It is 3-8 times more common in males than females (3).

Conservative treatment choices are limited in ulnar nerve entrapment neuropathy and very few studies about UNE, are available in literature. Among the evidence-based treatments the first choice is elbow splint (4). It is very important to avoid the movements that provoke the symptoms of UNE, the splint that is used in treatment allows the elbow to rest and lessens the inflammation and symptoms (4). During daytime elbow pads and/ or splints which keep the elbow in 30- 45 degree flexion position may be used (5-6). To prevent elbow flexion during sleep time a pillow /towel may be put on antecubital fossa or the elbow splint may be used during sleep time (4).

2-3 times a day the splint should be removed, and passive range of motion exercises should be performed. In a study it was found that using the splint at night does not only relieve the symptoms, but it also heals the ulnar nerve functions (7). On the other hand another study showed that using splint at night does not provide any additional benefit on avoiding symptom provoking positions (8).

Non-steroidal anti-inflammatory drugs (NSAID) are prescribed to relieve pain and inflammation in UNE. In case of there is no benefit of conservative treatment, when there is progressive paralysis in hand muscles and claw hand sign surgical treatment should be taken into consideration. Different surgical techniques are performed depending on the ulnar nerve entrapment region and elbow anatomy.

Conservative treatment choices of UNE are limited; since elbow splint limits daily living activities patient compliance is low and the results of elbow splint efficacy are controversial. While it was shown literaturally that physical medicine treatment modalities are effective in treatment of carpal tunnel syndrome (CTS) which is the most common upper extremity entrapment neuropathy (9, 10), there are a few studies about UNE treatment with physical medicine treatment modalities. It was shown in literature that continuous short-wave diathermy (SWD) application in CTS was effective on pain, function and symptom relief and this provided a basis for our study as CTS is an entrapment neuropathy similar to UNE. The aim of this study is researching the efficacy of SWD which is a deep heating modality in treatment of UNE. SWD is used either continuous or pulsed mode. Both thermal and non-thermal effects are seen due to absorption of electromagnetic energy in tissue. Among the thermal effects are; increase in blood flow, cell metabolism, tissue elasticity, changes in muscle relaxation and enzyme reactions due to increase in temperature. Superficial wound healing, decrease in edema, lymphedema, venous stasis ulcer are the result of non-thermal effects. Continuous SWD is used for the purpose of heating. It is essential to be precautious to avoid any kind of burn case. Pulsed-mode SWD is preferred for non-thermal effects although there is not enough evidence about its effects (11).

METHODS Patients and study design

The study was designed as randomized placebo controlled double blind research. 76 patients who applied İstanbul Fatih Sultan Mehmet Research and Training Hospital Physical Medicine and Rehabilitation clinic between February 2013- August 2013 and were diagnosed as UNE electrophysiologically according to criteria suggested by American Neurology Society were included into the study. 61 patients completed the study ( 1 patient continued the treatment in another hospital because of transportation, 3 patient left the treatment because of not being allowed by job boss, 4 patient left the treatment without giving any information, 7 patient completed the treatment but didn't come to the control examination). The hospital ethical committee permission was taken (FSMEAH-KAEK 2013/18 - 28.02.2013).

UNE Diagnosis Criteria suggested by American Neurology Society (12);

1. Ulnar nerve motor conduction velocity lower than 50 m/sec in elbow region
2. Elbow region ulnar nerve motor conduction velocity 10 m/sec lower than forearm region
3. More than 20% decrease in compound muscle action potential (CMAP) amplitude in above elbow stimulation compared to below elbow
4. Evident difference in configuration of above elbow CMAP compared to below elbow

If 2 of the criteria are positive it is a possible UNE diagnosis, and it is certain UNE diagnosis in case 3 criteria are positive.

Exclusion Criteria;

1. cervical radiculopathy
2. brachial plexopathy
3. ulnar nerve cut and trauma
4. sensation deficit in application region
5. diabetes mellitus
6. polyneuropathy
7. wound, burn, scar mark on forearm research region
8. presence of implant, prothesis, pin in tissue
9. not having well general health
10. epilepsy
11. presence of intrauterine device
12. presence of hearing instrument
13. presence of tumor, inflammatory states
14. pregnancy or pregnancy suspicion
15. being gotten radiotherapy ( during the last 6 months)

The patients were divided into two groups by coin toss randomization. The patients in the first group were applied continuous SWD treatment in 27.12 Hz frequency and for 20 minutes on elbow region by placing the elbow in 2 cm distance far from the condansator electrodes of SWD while the elbow is in 90 degree flexion. The second group patients were applied placebo SWD, the patients positioned same as the first group without turning on SWD. Both groups were given treatment 5 days a week and 10 session in total for two consecutive weeks. The physiotherapist that was applying the treatment on patients was not blind to treatment.

All patients were informed about UNE before the treatment, elbow positions and movements that might worsen the symptoms were being taught and recommended to avoid these positions, written consent was taken. The two group patients were prescribed elbow splint that keeps elbow in 30° flexion, to be used at night during the treatment period. Patient evaluation,before treatment, after treatment, first month after the treatment and third month after the treatment, was done by one physician (NBB) who was blind to all patients. The patients did not know if they were in treatment group or in control group until the study was completed.

The primary endpoint of this study is evaluation of pain intensity with VAS, secondary endpoint of this study is evaluation of changes in hypoesthesia and Tinel sign with quick-DASH, SF-36, dynamometer.

Assessments

In order to have a 15% relief in VAS there has to be 34 patients in each group according to power analysis. The study was designed with 76 patients, because of some of the volunteers not completing the treatment, 31 patients participate in treatment group and 30 patients participate in control group, as a total studt was completed with 61 patients.

The age, height, weight, gender, occupation, education level, dominant hand, affected extremity, history of repetitive trauma of patients were recorded. BMI (body mass index) has been calculated by using the data of height and weight with the formula of BMI= body mass (kg)/ (height)² (m²). The patients with BMI > 30 were accepted as obese.

The patients were evaluated by physical examination, daily living activities, pain and grip strength before treatment, after treatment, one month after treatment and three months after treatment. In order to evaluate the patients Visiual Analogue Scale (VAS), Short Form 36, Quick -DASH, muscle assessment scale, grip strength with dynamometer used, and if it was present of claw hand deformity, hypothenar atrophy, Tinel sign, hypoesthesia (thenar/ hypothenar), Froment sign, Wartenberg sign recorded. McGowen classification has been performed before treatment.

Statistical analysis For statistical analysis NCSS (Number Cruncher Statistical System) 2007&PASS (Power Analysis and Sample Size) 2008 Statistical Software (Utah, USA) softwares were used. Besides descriptive statistical methods ( mean, standard deviation, median, frequency, rate, minimum, maximum), for comparison of quantitative data between two groups; if parameters were normally distributed student t test, if they were not normally distributed Mann Whitney U test were used. To compare qualitative data Fisher's exact test and Yates Continuity Corection Test (Yates Corected chi-square) were used. For in-group analysis in follow-ups; comparison of normally distributed parameters were done by paired samples Test, and Wilcoxon Signed Ranks Test was preferred for parameters that were not normally distributed. Statistical significance was measured with p<0,01 and p<0,05.

DISCUSSION

UNE is an upper extremity disease which is second most common peripheral neuropathy after CTS, that causes functional insufficiency in daily living activities and praxis requiring works and therefore results in work loss. The main goal in UNE treatment is; increasing the life quality in the long term by relieving the symptoms, lessening the compression on the nerve, preventing the nerve damage, stopping the present nerve damage, preservation of physical function and social participation.

Although UNE is the second most common peripheral neuropathy there is no consensus about its treatment according to currently present studies. The present treatment options are divided into two as; conservative treatment and surgery. Conservative treatment option is composed of; patient education, exercise, splinting, physical medicine modalities, pharmacological treatments. In case there is no enough clinical relief in conservatively treated patients, surgery is preferred. In a study was made by Hong et al; 10 patients ( 12 ulnar nerve neuropathy cases) were divided into two groups. Group A which was composed of 5 cases were given an elbow splint that keeps elbow in 30-35° flexion position, group B which was composed of 7 cases were given splint and administered single dose of 40 mg triamsinolone injection in elbow near ulnar nerve (6). In first month control examination there was an increase in nerve conduction velocity of group A, there was same amount increase in both group A and group B in sixth month control examination. Svernlöv et al. studied 51 UNE patients by dividing them into 3 groups (13). Group 1 was given splint and recommended to avoid symptom provoking activities, group 2 was given nerve gliding exercises and recommended to avoid symptom provoking activities, group 3 was recommended only to avoid symptom provoking activities. It was found that splint and nerve gliding exercises did not provide any additional benefit on clinical outcome. In our study we recommend every patient elbow splint that keeps elbow in 30° flexion. Despite some studies showing the night splint is beneficial, some other studies show that it has no effect on clinical outcome.

In a study of Nakamichi et al. 77 patients ( 80 ulnar neuropathy cases) were told to avoid positions that causes mechanical pressure on ulnar nerve (14). The cases that had relief in complaints were followed up until 1 year. It was concluded that mild and moderate cases of UNE could be treated b avoiding smptom provoking activities compared to severe cases. According to our study; the similar improvement in VAS, quick-DASH, dynamometer, SF-36 results were related to avoidance of symptom provoking activites.

In a study made by Özkan et al., 32 cases of UNE were divided into two groups and first group was given ultrasound treatment, second group was given low level laser treatment for 2 weeks, 5 days per week (15). It was found that there was clinical and electrophysiological improvement in both groups in first month control examination and there was no significant difference between groups. Guiseppina et al. divided 22 patients (34 cases) of CTS into two equal groups, and studied effect of deep heating modality (7). First group was treated 20 minutes per session, 2 session per week with a microwave energy producing physical therapy modality and in total 6 sessions of treatment were given. Second group was placebo treatment group, was given same duration and same times sham treatment. It was found that deep heating had a significant effect on pain and function compared to placebo group. İncebıyık et al. studied effect of SWD on 31 patients (58 cases) of mild or moderate CTS dividing into two groups (16). The treatment was designed as 5 sessions per week, 15 sessions in total. First group was given superficial heating treatment, SWD, nerve and tendon gliding exercises, second group was given superficial heat treatment, placebo SWD, nerve and tendon gliding exercises. It was found that SWD was effective in CTS on pain, function, clinical symptoms improvement. We studied effectiveness of SWD, which is a deep heating modality similar to US, microwave, by controlling with a placebo group. Because of having a few studies about UNE and small sample sizes there are different results about deep heating effectiveness.

Our study is important because of being randomized placebo controlled double blind, getting patients evaluated in many aspects, being the first studying SWD effectiveness on UNE. Having a small sample size and short follow up period are limitations of our study. Because of not having many studies about SWD effectiveness in UNE treatment, the session number was decided depending on the clinical experiences which is another limitation of our study. In our opinion; it will be useful to show the effect of physical medicine modalities in UNE treatment with studies which are planned with more patients, more sessions and longer period of follow ups with different physical medicine modalities which are organized as placebo controlled.

Financial Support There was no any support from any foundation or settlement. The patients were not paid for volunteering the study.

ELIGIBILITY:
Inclusion Criteria:

* UNE Diagnosis Criteria suggested by American Neurology Society (12);

  1. Ulnar nerve motor conduction velocity lower than 50 m/sec in elbow region
  2. Elbow region ulnar nerve motor conduction velocity 10 m/sec lower than forearm region
  3. More than 20% decrease in compound muscle action potential (CMAP) amplitude in above elbow stimulation compared to below elbow
  4. Evident difference in configuration of above elbow CMAP compared to below elbow

     If 2 of the criteria are positive it is a possible UNE diagnosis, and it is certain UNE diagnosis in case 3 criteria are positive.

     Exclusion Criteria:

  <!-- -->

  1. cervical radiculopathy
  2. brachial plexopathy
  3. ulnar nerve cut and trauma
  4. sensation deficit in application region
  5. diabetes mellitus
  6. polyneuropathy
  7. wound, burn, scar mark on forearm research region
  8. presence of implant, prothesis, pin in tissue
  9. not having well general health
  10. epilepsy
  11. presence of intrauterine device
  12. presence of hearing instrument
  13. presence of tumor, inflammatory states
  14. pregnancy or suspect of pregnancy
  15. being exposed to radiotherapy ( during the last 6 months)

Ages: 16 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2013-08-31 (Actual)

PRIMARY OUTCOMES:
pain in hand and elbow due to ulnar nerve entrapment | 3 months
  the pain of the participants were measured with VAS (visiual analogy scale). the difference between pain in baseline and 3 months after treatment were compared in order to get the primary outcome measure
hand function in daily living activities | 3 months
  the progress in function was measured with quick -DASH questionnaire. the baseline measure and 3 months after treatment measures were compared in order to get the primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: naciye bilgin badur, doctor, Principal Investigator — sureyyapasa chest diseases and chest surgery hospital
Locations (1):
- Sureyyapasa Chest Diseases and Chest Surgery Hospital, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
statistical analysis and study method and design will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: as soon as the article is pressed as long as the article is in press
Access Criteria: via article

REFERENCES:
- [Result] 1.Özçete Z.A, On A.Y. : Ulnar sinir tuzak nöropatileri. TürkFiz Tıp Rehab Derg. 56; 190-5, 2010 2. Robertson C, Saratsiotis J. A review of compressive ulnar neuropathy at the elbow. J Manipulative Physiol Ther 2005;28:345. 3. Piligian G, Herbert R, Hearns M, Dropkin J, Landsbergis P, Cherniack M. Evaluation and management of chronic workrelated musculoskeletal disorders of the distal upper extremity. Am J Ind Med 2000;37:75-93. 4. Sailer SM. The role of splinting and rehabilitation in the treatment of carpal and cubital tunnel syndromes. Hand Clin 1996;12:223-41. 5. Seror P. Nocturnal orthosis: a new treatment of compression of the ulnar nerve at the elbow. 30 cases. Rev Neurol (Paris). 1994 Oct;150(10):721-7. 6. Hong CZ, Long HA, Kanakamedala RV, Chang YM, Yates L. Splinting and local steroid injection for the treatment of ulnar neuropathy at the elbow: clinical and electrophysiological evaluation. Arch Phys Med Rehabil 1996;77:573-7. 7. Frasca G, Maggi L, Padua L, Ferrara PE, Granata G, Minciotti I, Marzetti E, Specchia A, Ronconi G, Rabini A, Bertolini C, Piazzini DB. Short-term effects of local microwave hyperthermia on pain and function in patients with mild to moderate carpal tunnel syndrome: a double blind randomized sham-controlled trial. Clin Rehabil. 2011 Dec;25(12):1109-18. Epub 2011 Sep 21. 8. Svernlöv B, Larsson M, Rehn K, Adolfsson L. Conservative treatment of the cubital tunnel syndrome. J Hand Surg Eur Vol 2009;34:201. 9. Zlowodzki M, Chan S, Bhandari M, et al. Anterior transposition compared with simple decompression for treatment of cubital tunnel syndrome. A meta-analysis of randomized, controlled trials. J Bone Joint Surg Am. 2007;89(12):2591-2598. 10. Gay JR, Love JG. Diagnosis and treatment of tardy paralysis of the ulnar nerve; based on a study of 100 cases. J Bone Joint Surg Am. 1947;29(4):1087-1097. 11. Jeffrey R. Basford, G. David Baxter. Therapeutic Physical Agents. Walter R. Frontera, Joel A. DeLisa( Eds.). Physical Medicine & Rehabilitation. 5. ed. Philadelphia: Lippincott Williams & Wilkins;2010 :1698-1700 12. Campbell WW. Guidelines in electrodiagnostic medicine. Practice parameter for electrodiagnostic studies in ulnar neuropathy at the elbow. Muscle Nerve Suppl 1999;8:S171-205. [Abstract] 13.Svernlöv B, Larsson M, Rehn K, Adolfsson L. Conservative treatment of the cubital tunnel syndrome. J Hand Surg Eur Vol 2009; 34:201. 14. Nakamichi K, Tachibana S, Ida M, Yamamoto S (2009) Patient education for the treatment of ulnar neuropathy at the elbow. Arch Phys Med Rehabil 90:1839-1845 15. Ozkan FU, Saygı EK, Senol S, Kapcı S, Aydeniz B, Aktas I, Gozke E. New treatment alternatives in the ulnar neuropathy at the elbow: ultrasound and low-level laser therapy. Acta Neurol Belg DOI 10.1007/s13760-014-0377-9 16. Incebiyik S, Boyaci A, Tutoglu A. Short-term effectiveness of short-wave diathermy treatment on pain, clinical symptoms, and hand function in patients with mild or moderate idiopathic carpal tunnel syndrome. J Back Musculoskelet Rehabil. 2014 Jul 24. [Epub ahead of print]